CLINICAL TRIAL: NCT00003853
Title: Phase II Trial of 4'-IODO-4'-Deoxydoxorubicin in Primary Amyloidosis (AL)
Brief Title: 4'-Iodo-4'-Deoxydoxorubicin in Treating Patients With Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Morie Abraham Gertz, M.D., Mayo Clinic
Purpose: Treatment
Other Study IDs: CDR0000067016; P30CA015083 (NIH); 988003 (Other: Mayo Clinic Cancer Center); T98-0003 (Other: NCI Protocol); 302-99 (Other: Mayo Clinic IRB)
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — 4'-deoxy-4'-iododoxorubicin

INTERVENTIONS:
Drug: 4'-iodo-4'-deoxydoxorubicin

SUMMARY:
RATIONALE: 4'-Iodo-4'-deoxydoxorubicin may improve organ dysfunction and ease symptoms caused by primary systemic amyloidosis.

PURPOSE: Phase II trial to study the effectiveness of 4'-iodo-4'-deoxydoxorubicin in treating patients who have primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the clinical efficacy of 4'-iodo-4'-deoxydoxorubicin in producing palliation of symptoms and/or improvement of organ dysfunction caused by organ infiltration by amyloid in patients with primary systemic amyloidosis. II. Assess the safety profile, with emphasis on cardiac safety, of this drug in these patients. III. Evaluate the time to progression of amyloidosis-associated clinical symptoms and/or organ dysfunction, duration of response, and survival of these patients on this regimen.

OUTLINE: Patients receive 4'-iodo-4'-deoxydoxorubicin IV over 1 hour once a week for 4 weeks. Courses are repeated every 12 weeks. Treatment continues for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histochemically proven primary systemic amyloidosis (AL) No presence of non-AL amyloidosis No amyloid-specific syndrome (e.g., skin purpura or carpal tunnel syndrome) as only evidence of disease No vascular amyloid only in a bone marrow biopsy specimen or in a plasmacytoma Must have symptomatic organ involvement with amyloid (e.g., liver, mild cardiac, renal, or soft tissue involvement, or grade 1 or 2 peripheral neuropathy) Demonstrable M-protein in the serum/urine OR Clonal population of plasma cells in the bone marrow OR Immunohistochemical stain with anti-light chain antisera of amyloid fibrils No clinically overt multiple myeloma (i.e., monoclonal BMPC greater than 20% and at least one of the following: bone lesions, anemia, or hypercalcemia)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Total bilirubin less than 2.0 mg/dL OR Direct bilirubin no greater than 1.0 mg/dL Alkaline phosphatase no greater than 4 times upper limit of normal (ULN) ALT or AST no greater than 3 times ULN Renal: Creatinine clearance greater than 40 mL/min Cardiovascular: Echocardiographic ejection fraction greater than 50% At least 3 years since prior enzyme documented myocardial infarction Interventricular septal thickness no greater than 20 mm No New York Heart Association class III or IV heart failure No grade 2 or 3 A-V block No chronic atrial fibrillation No sustained (greater than 30 seconds) ventricular tachycardia or frequent episodes (greater than 20 in 24 hours) of nonsustained ventricular tachycardia or ventricular pairs, detected by 24-hour ambulatory electrocardiographic monitoring Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV positive allowed No uncontrolled infection No severe diarrhea not controllable with medication or that requires total parenteral nutrition No other concurrent active malignancy except nonmelanoma skin cancer or cervical cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 weeks since prior interferon alfa Chemotherapy: No prior anthracyclines greater than 120 mg/m2 At least 6 weeks since prior melphalan or other alkylating agents Endocrine therapy: At least 6 weeks since prior high dose dexamethasone Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 1999-04; Primary Completion 2000-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morie A. Gertz, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mayo Clinic Cancer Center, Rochester, Minnesota
- University of Pavia, Pavia, Italy

REFERENCES:
- [Result] Gertz MA, Lacy MQ, Dispenzieri A, Cheson BD, Barlogie B, Kyle RA, Palladini G, Geyer SM, Merlini G. A multicenter phase II trial of 4'-iodo-4'deoxydoxorubicin (IDOX) in primary amyloidosis (AL). Amyloid. 2002 Mar;9(1):24-30. doi: 10.3109/13506120209072441. PMID 12000194